CLINICAL TRIAL: NCT05851664
Title: Do we Intubate Faster With the Videolaryngoscope?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mongi Slim Hospital (Other)
Responsible Party: Principal Investigator, Mhamed Sami Mebazaa, Professor, Mongi Slim Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Time to intubate VL
Record Dates: First submitted 2023-04-30; First posted 2023-05-10 (Actual); Last update posted 2023-05-23 (Actual); Status verified 2023-05

CONDITIONS: Laryngoscopy; General Anesthesia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group Direct laryngoscopy (DL) (Active Comparator): Group DL: intubated with direct laryngoscopy type Macintosh.
  Interventions: Device: intubation by direct laryngoscopy
- Group vidéo Laryngoscopy (VL) (Experimental): Group VL: intubated with a video laryngoscope type McGrath
  Interventions: Device: Intubation by videolaryngoscopy

INTERVENTIONS:
Device: intubation by direct laryngoscopy — intubation using a direct laryngoscopy type macintosh
  Other Names: DL
  Arms: Group Direct laryngoscopy (DL)
Device: Intubation by videolaryngoscopy — Intubation using a videolaryngoscope type McGrath
  Other Names: VL
  Arms: Group vidéo Laryngoscopy (VL)

SUMMARY:
The Aim of the study was to determine the impact of the videolaryngoscpe on the time needed to intubate.

This was a Prospective, randomized, simple blinded study. The participants intubated patients for surgery under general anesthesia either with direct laryngoscpy or with videolaryngoscopy.

DETAILED DESCRIPTION:
Intubation on full stomach is at high risk of pulmonary suction. It must be quick, as this risk increases with the time needed to intubate. Videolaryngoscope (VL) is recommended in case of difficult airway. Yet, its interest in full stomach remains unclear, as the time needed to intubate with a VL is variable in literature. The Aim of the study was to determine the impact of the videolaryngoscpe on the time needed to intubate.

This was a Prospective, randomized, simple blinded study. The participants intubated patients for surgery under general anesthesia either with direct laryngoscpy or with videolaryngoscopy.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years-old;
* ASA status 1 to 3;
* General anesthesia and intubation.

Exclusion Criteria:

* Difficult intubations criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
Time needed to intubate | during the intubation
  Time needed to the operator to pass the tube through vocal cords in seconds

SECONDARY OUTCOMES:
Difficulty of the laryngoscopy | at the end of intubation
  cormack anf lehane grade (1 to 4) 1 and 2 indicate easy laryngoscopy and 3 and 4 indicate difficult laryngoscopy
Number of intubation attempts. | at the end of intubation
  number of attempts needed to intubate
Major desaturation | during intubation
  an oximetry under 90 %

CONTACTS AND LOCATIONS:
Overall Officials: Mhamed Sami MS Mebazaa, Pr, Principal Investigator — Mongi Slim Hospital
Locations (1):
- Mongi Slim hospital, Tunis, Tunisia

IPD SHARING:
Plan to Share IPD: No